CLINICAL TRIAL: NCT05021588
Title: Challenges in Steroid and Anticoagulant Therapy in Severe COVID-19 Pneumonia: A Prospective Study
Brief Title: Steroid and Anticoagulant Therapy in covid19
Acronym: SARS-CoV-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa mahmoud Abd El Rady, lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: anticoagulant in covid19
Record Dates: First submitted 2021-08-16; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Pneumonia, Viral
MeSH Terms: conditions — Pneumonia, Viral | interventions — Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A:dexamethasone (Experimental)
  Interventions: Procedure: steroid and anticoagulants according to different protocols.
- Group B: prednisolone or methyl prednisolone according to D-dimer levels. (Experimental)
  Interventions: Procedure: steroid and anticoagulants according to different protocols.
- Group C: prednisolone or methylprednisolone and anticoagulants according to the flexible protocol. (Experimental)
  Interventions: Procedure: steroid and anticoagulants according to different protocols.

INTERVENTIONS:
Procedure: steroid and anticoagulants according to different protocols. — As no standard treatment for COVID-19 was approved; there are many treatment protocols for anti-inflammatory corticosteroids and anti-coagulantsfor severe COVID-19 pneumonia cases, this study aims to assess the most suitable modality in this high-risk group.

SUMMARY:
As COVID-19 has neither standard treatment protocol nor guidelines, there are many treatment protocols foranti-inflammatory corticosteroids and anti-coagulations for severe COVID-19 pneumonia patients. This study aimed to assess the most suitable modality in this high-risk group.

Methods: A prospective, experimental study design was adopted, that included 123 severe COVID-19 pneumonia patientsadmitted at Assiut UniversityHospital from April 10th, 2020, to September10th, 2020. Patients were divided into 3 groups according to a combined corticosteroid and anticoagulants therapy protocols. Group A included 32 patients, group B included 45 patients, and group C included 46 patients. Assessment of cases was conducted according to the treatment type and duration, weaning duration from oxygen therapy, length of hospital and ICU stay, and complications during treatment.Three months follow up after discharge was performed.

ELIGIBILITY:
Inclusion Criteria:

* respiratory distress [respiratory rate (RR) >30 breaths/min at rest], mean oxygen saturation ≤93%,ratio of arterial oxygen partial pressure to fractional inspired oxygen (PaO2/FiO2) ≤300 mmHg,>50% lung involvement on imaging within 24 to 48 hours of admission

Exclusion Criteria:

* pnumonia not caused by covid19

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-08-02 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Outcome of patients after corticosteroids and anti-coagulants for severe COVID-19 pneumonia | 5 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marwarady, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No